CLINICAL TRIAL: NCT02028390
Title: Scout Overlay-Trace-On-Thermal Feature in a Wound Clinic Setting: A Prospective Study
Brief Title: Overlaying a Visual Wound Trace Onto Its Thermal Image in a Wound Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wound Vision (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: WV13CL-0008 Revision 02
Record Dates: First submitted 2013-12-23; First posted 2014-01-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Wounds and Injuries
Keywords: wounds; thermal; temperature; periwound; camera; imaging
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subjects with external wounds (Experimental): Subjects with external wounds or body surface areas of interest are imaged visually and thermally with the Scout to trace the wound's perimeter visually and measure thermal variation data as described in the primary outcomes, using the ImageReview software.
  Interventions: Device: Scout takes visual and thermal images of external wounds; Device: ImageReview's visual perimeter trace of the external wound; Device: ImageReview's External Wound Trace Overlay; Device: ImageReview's unaffected reference area selected; Device: Adjacent tissue trace of the wound trace overlay

INTERVENTIONS:
Device: Scout takes visual and thermal images of external wounds — All images are taken after the wound has acclimated.
  Other Names: Wound Measuring and Monitoring System/WMMS (past)
Device: ImageReview's visual perimeter trace of the external wound — Trace is drawn by the study staff using the ImageReview software.
Device: ImageReview's External Wound Trace Overlay — Study staff overlay the trace of the visual external wound's perimeter onto the corresponding thermal image of the external wound.
Device: ImageReview's unaffected reference area selected — Study Staff select an unaffected reference area of an adjacent body surface.
Device: Adjacent tissue trace of the wound trace overlay — Study staff select an adjacent tissue trace of the wound trace overlay

SUMMARY:
The purpose of this study is to test and evaluate how well a medical imaging device that takes both visual and thermal pictures of wounds or body surface areas of interest can help collect added information about the wounds or body surface areas of interest in a wound clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater, of either gender and of any ethnic background
* Able to tolerate position change(s) and turns for up to 10 minutes comfortably
* Have an existing external wound or body surface area of interest:

  * External wound or body surface area of interest must be in separate body locations (ex: one on the right heel, one on the left heel, and the other on the sacrum)
* Have qualifying external wound or body surface area of interest:

  * External wound or body surface area of interest that fits entirely within the field of view and does not wrap around a body edge
  * No device or treatment will obscure the external wound or body surface area of interest

Exclusion Criteria:

* Neonatal and pediatric patients
* Pregnant women
* Cannot tolerate position changes for up to 10 minutes comfortably (per external wound site imaged)
* On therapies or treatments which cannot be safely suspended long enough to conduct an imaging session as determined by facility policy
* Have a wound dressing or medical device which cannot or should not be removed as determined by site investigator
* Have an external wound with excessive or heavy exudate that cannot be controlled during the imaging session. Excessive drainage can obscure external wound features.
* If the patient has a complex external wound:

  * The external wound wraps around a body edge or otherwise cannot be imaged entirely within the visual field of view.
  * From visual assessment, the external wound edges are not definable and/or cannot be clearly distinguished from other conditions near external wound (E.g. breakdown or the deterioration of the surrounding body surfaces due to other conditions such as cancer or other types of ulcers makes determining the edge of the external wound impossible).
* Have not provided signed informed consent
* Non-English speaking
* Subjects in isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pixel gradient of the thermal wound surface | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Pixel gradient of the thermal wound surface will be measured, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Mean pixel value of the thermal wound surface | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Mean pixel value of the thermal wound surface will be measured, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Mode pixel value of the thermal wound surface | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Mode pixel value of the thermal wound surface will be measured, with changes documented during regularly scheduled wound care visits at the wound clinic for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Pixel gradient of the thermal unaffected area of body surface selected | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Pixel gradient of the the thermal unaffected area of body surface selected will be measured, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Highest pixel value of the thermal wound surface | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Highest pixel value of the thermal wound surface will be measured, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Lowest pixel value of the thermal wound surface | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Lowest pixel value of the thermal wound surface will be measured, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Comparison of adjacent tissue trace around the wound bed's surface's relative temperature (Centigrade and Fahrenheit) to the unaffected reference area's relative temperature (Centigrade and Fahrenheit). | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Comparison of adjacent tissue trace around the wound bed's surface's relative temperature (Centigrade and Fahrenheit) to the unaffected reference area's relative temperature (Centigrade and Fahrenheit), with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Comparison of wound surface's relative temperature (Centigrade and Fahrenheit) to the unaffected reference area's relative temperature (Centigrade and Fahrenheit). | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Comparison of wound surface's relative temperature (Centigrade and Fahrenheit) to the unaffected reference area's relative temperature (Centigrade and Fahrenheit), with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Wound surface's % relative temperature above, below, or equal to the unaffected reference area's temperature | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Wound surface's % relative temperature above, below, or equal to the unaffected reference area's relative temperature, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.
Adjacent tissue trace's surface % relative temperature above, below, or equal to the unaffected reference area's temperature | Weeks 1-104, with week 104 as an estimated time frame maximum, for which changes will be measured and documented
  Adjacent tissue trace's surface's % relative temperature above, below, or equal to the unaffected reference area's relative temperature, with changes documented during regularly scheduled wound care visits for a minimum of two visits and may continue at the discretion of the primary investigator and the subject until the subject no longer qualifies or the study is ended, when 100 subjects are enrolled or the study has completed two years.

CONTACTS AND LOCATIONS:
Overall Officials: Aletha W. Tippett, M.D., Principal Investigator — Integrative Center for Healing
Locations (1):
- Integrative Center for Healing, Cincinnati, Ohio, United States